CLINICAL TRIAL: NCT06924931
Title: Five-year Recurrence and Postoperative Complications After Laparoscopic Complete Mesocolic Excision- a Population-Based, Multicentred Study
Brief Title: Five-year Recurrence After LCME
Status: Completed | Type: Observational
Sponsor: Gødstrup Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LapCMEinCDR
Record Dates: First submitted 2025-04-05; First posted 2025-04-13 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-04

CONDITIONS: Colon Cancer Stage I; Colon Cancer Stage II; Colon Cancer Stage III
Keywords: colon cancer; LCME; CME; recurrence; laparoscopic complete mesoclic excision
MeSH Terms: conditions — Colonic Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PRE: pre-implementation group
- POST: post-implementation group
  Interventions: Behavioral: LCME training programme

INTERVENTIONS:
Behavioral: LCME training programme — A LCME training program was conducted from March 2017 to October 2017 in the CDR, inspired by the National English Laparoscopic Colorectal Surgery Course. All certified colorectal surgeons from three public hospitals in the CDR were invited. The training programme was conducted over 2-3 days, occurring twice within an 8-month period.
  Groups: POST

SUMMARY:
A register-based study is conducted to examine clinical outcomes following a population-based, multi-centred implementation of Laparoscopic Complete Mesocolic Excision (LCME) in the Central Denmark Region, Denmark.

DETAILED DESCRIPTION:
This study was conducted as a population-based "before-and-after" cohort study following the implementation of LCME in the Central Denmark Region (CDR), Denmark, in 2017. The IDEAL framework (Idea, Development, Evaluation, Assessment, Long-term) was used for examining the outcome of a training program on the LCME adoption.

Training programme A LCME training program was conducted from March 2017 to October 2017 in the CDR, inspired by the National English Laparoscopic Colorectal Surgery Course.

Patients This study included all colon cancer patients undergoing a curative-intent bowel resection in the defined timeframe. Exclusion criteria comprised: 1) another synchronous colon cancer; 2) metastatic disease at the time of surgery; 3) non-curative procedures or local resections only; 4) Danish residency <10 years preoperatively; and 5) non-colon primary cancer.

Data sources The DCCG database, a national registry of newly diagnosed colon cancer patients, was used to identify the primary cohort. For follow-up data beyond 30 days after surgery, the cohort was linked to the following registries: 1) the Danish Civil Registration System (DCRS), 2) the Danish Cancer Registry (DCR), 3) the Danish National Patient Registry (DNPR), 4) the Danish Pathology Registry (DPR) and the Danish Pathological Data Bank (DPDB).

Outcome The primary outcome was the cumulative incidence of colon cancer recurrence 5 years after surgery. A validated algorithm was used to identify recurrence.

The secondary outcome was postoperative complications within 30 days graded by the Clavien- Dindo Classification (CDC) (minor: I-II, major: III-V).

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed colon cancer patients.

Exclusion Criteria:

1. another synchronous colon cancer
2. metastatic disease at the time of surgery
3. non-curative procedures or local resections only
4. Danish residency <10 years preoperatively
5. non-colon primary cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study included all colon cancer patients undergoing a curative-intent bowel resection in Central Denmark Region, Denmark in the following timeframe: (January 1, 2015-December 31, 2016) and (January 1, 2018-December 31, 2019).
Sampling Method: Non-Probability Sample
Enrollment: 2529 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Recurrence | From surgery to date of recurrence or end of 5-years follow up.
  The cumulative incidence of colon cancer recurrence 5 years after surgery.

SECONDARY OUTCOMES:
mortality | From surgery to the date of mortality or end of 5-years follow-up.
  The cumulative incidence of mortality 5 years after surgery.
postoperative complications | 30 days after primary surgery
  30-day postoperative complications

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared as this is a register-based study, and according to the GLPR and Danish law, the IPD date cannot be shared.